CLINICAL TRIAL: NCT06089369
Title: Postoperative Adjuvant Sintilimab in Hepatocellular Carcinoma With Microvascular Invasion: A Multicenter, Phase III, Randomized Study
Brief Title: Postoperative Adjuvant Sintilimab in Hepatocellular Carcinoma With Microvascular Invasion
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Chen Xiaoping, Professor, Tongji Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Adjuvant-01
Record Dates: First submitted 2023-10-13; First posted 2023-10-18 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Hepatocellular Carcinoma
Keywords: Programmed Cell Death 1; Checkpoint Inhibitor; Immunotherapy; Adjuvant; Hepatocellular Carcinoma; Microvascular Invasion
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — sintilimab; Watchful Waiting

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sintilimab for six months group (9 cycles) (Experimental): Patients receive Sintilimab at a dose of 200 mg via intravenous injection, with one cycle every three weeks, for a total of 9 cycles or until disease recurrence or intolerable adverse effects occurred.
  Interventions: Drug: Sintilimab (9 cycles)
- Sintilimab for one year group (18 cycles) (Experimental): Patients receive Sintilimab at a dose of 200 mg via intravenous injection, with one cycle every three weeks, for a total of 18 cycles or until disease recurrence or intolerable adverse effects occurred.
  Interventions: Drug: Sintilimab (18 cycles)
- Active surveillance (Active Comparator): Patients are closely monitored postoperatively.
  Interventions: Other: Active surveillance

INTERVENTIONS:
Drug: Sintilimab (9 cycles) — IV infusion of Sintilimab （200mg intravenously every 3 weeks for a total of 9 cycles）
  Other Names: IBI 308
  Arms: Sintilimab for six months group (9 cycles)
Drug: Sintilimab (18 cycles) — IV infusion of Sintilimab （200mg intravenously every 3 weeks for a total of 18 cycles）
  Other Names: IBI 308
  Arms: Sintilimab for one year group (18 cycles)
Other: Active surveillance — Active surveillance
  Arms: Active surveillance

SUMMARY:
To compare the impact on recurrence risk of adjuvant Sintilimab (a recombinant fully human anti-PD-1 monoclonal antibody) for patients with hepatocellular carcinoma and microvascular invasion (MVI) after hepatectomy.

DETAILED DESCRIPTION:
This study is a prospective, multicenter, open-label, randomized controlled clinical trial, aiming to recruit 360 patients with MVI-positive HCC who have undergone surgical resection. The patients will be randomly divided into three groups: the first group will receive six months of adjuvant therapy with Sintilimab (200 mg every three weeks for a total of 9 cycles), the second group will receive one year of adjuvant therapy with Sintilimab (200 mg every three weeks for a total of 18 cycles), and the Active surveillance group will be closely followed postoperatively. A maximum of one postoperative adjuvant TACE is permitted.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a histopathological diagnosis of HCC
* Undergone a curative resection
* Pathologically confirmed HCC with microvascular invasion (MVI)
* Aged 18-75 years
* No previous systematic treatment and locoregional therapy for HCC prior to randomization
* Absence of major macrovascular invasion
* No extrahepatic spread
* Full recovery from Curative resection within 4 weeks prior to randomization
* Child-Pugh: Grade A or B(7)
* ECOG-PS score: 0 or 1
* Subjects with HCV- RNA (+) must receive antiviral therapy
* Adequate organ function

Exclusion Criteria:

* Known fibrolamellar HCC, sarcomatoid HCC, mixed cholangiocarcinom or recurrent HCC
* Any preoperative treatment for HCC including local and systemic therapy
* Have received more than 1 cycle of adjuvant TACE following surgical resection
* Any acute active infectious diseases, active or history of autoimmune disease, or immune deficiency
* Known history of serious allergy to any monoclonal antibody or targeted anti-angiogenic drug
* Subjects with inadequately controlled hypertension or history of hypertensive crisis or hypertensive encephalopathy
* Cardiac clinical symptom or cardiovascular disease that is not well controlled
* Thrombosis or thromboembolic event within 6 months prior to the start of study treatment
* Any persistent serious surgery-related complications; esophageal and/or gastric variceal bleeding within 6 months
* Abdominal fistula, gastrointestinal perforation or intraperitoneal abscess within 6 months prior to the start of study treatment
* Inability or refusal to comply with the treatment and monitoring

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Recurrence-Free Survival (RFS) | Randomization up to 60 months
  RFS is defined as the time from randomization to the first documented occurrence of local, regional, or metastatic HCC as determined by BIRC, or death from any cause (whichever occurs first).

SECONDARY OUTCOMES:
RFS Rate at 12 ,24 , 36 , 60 Months | Randomization up to 60 months
  RFS is defined as the time from randomization to the first documented occurrence of local, regional, or metastatic HCC as determined by BIRC, or death from any cause (whichever occurs first).
Overall Survival (OS) | Randomization up to 60 months
  OS is defined as the time from randomization to death from any cause
Adverse events | Baseline up to 60 months
  The incidence and severity of adverse events (AEs) and serious adverse events (SAEs) as assessed by CTCAE v5.0
Quality of Life (QoL) Scale Score | Baseline up to 60 months
  Change from Baseline in European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Core 30 (QLQ-C30) and Hepatocellular Carcinoma Module (EORTC QLQ-HCC18) Scale Score

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China